CLINICAL TRIAL: NCT00338806
Title: Prevention for Symptomatic Offspring of Bipolar Parents
Brief Title: Early Detection and Prevention of Mood Disorders in Children of Parents With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #5067; K23MH071530 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Bipolar Disorder; Depression
Keywords: Prevention; Mood Disorders; Unipolar Depression
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders; Depressive Disorder | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpersonal Psychotherapy-Prevention (Experimental): Participants will receive interpersonal psychotherapy for prevention with adolescents
  Interventions: Behavioral: Interpersonal psychotherapy for prevention with adolescents
- Educational and Clinical Monitoring (Active Comparator): Participants will receive educational clinical monitoring
  Interventions: Behavioral: Educational clinical monitoring

INTERVENTIONS:
Behavioral: Interpersonal psychotherapy for prevention with adolescents — Individual interpersonal psychotherapy with the adolescents will be conducted over 12 weeks and will include a family psychoeducation component.
  Other Names: IPT-PA
  Arms: Interpersonal Psychotherapy-Prevention
Behavioral: Educational clinical monitoring — Educational clinical monitoring will include two individual sessions of psychoeducation on mood disorders with the adolescent followed by monthly (and if needed bimonthly) meetings with therapist. If more sessions are required, a referral will be made.
  Other Names: ECM
  Arms: Educational and Clinical Monitoring

SUMMARY:
This study will develop strategies for early detection and prevention of mood disorders and associated impairment in adolescent children of parents with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar Disorder (BD) is a serious medical illness that causes drastic shifts in a person's mood, energy, and ability to function. BD symptoms alternate from increased energy, restlessness, and overly good mood to a lasting sad, anxious, or empty mood and feelings of hopelessness or pessimism. Research suggests that children of parents with BD are at risk for developing mood disorders because of predisposing genetic factors and stressful life events, many of which may be related to their parents' unstable clinical state. Adolescent children of parents with BD must deal simultaneously with the difficult task of negotiating their own developmental transitions, as well as living with a parent with BD. It may be possible to detect symptoms of BD or other mood disorders early in adolescence and prevent the disorder from further interfering with someone's life. This study will develop and refine strategies for early detection and primary prevention of mood disorders and associated impairment in adolescent children of parents with BD.

Participants in this single-blind study will be randomly assigned to receive either interpersonal psychotherapy with adolescents (IPT-PA) or a control intervention, educational clinical monitoring (ECM), for 12 weeks. Participants assigned to IPT-PA will attend twelve sessions. The first four sessions will last 90 minutes each, and will include both family psychoeducation and individual psychotherapy with the adolescent. The remaining sessions will be 45 minutes each, and will include only individual psychotherapy with the adolescent. Participants assigned to ECM will each be assigned to a therapist. During the initial two sessions, which will take place over 2 consecutive weeks, the therapist will focus on mood disorder psychoeducation and participants will receive related written educational material. Participants will then meet with their therapists monthly for 30-minute sessions. Symptoms and functioning will be assessed, but no assistance on building interpersonal skills will be provided. A participant may request a second session each month, but if more than two monthly sessions are required, the participant will be referred for therapy. Mood episodes and symptoms, symptom severity, and functioning will be assessed for all participants at Weeks 6 and 12 and Months 6, 12, and 18 post-treatment.

ELIGIBILITY:
Inclusion Criteria for Parents:

* Diagnosis of BD I or II
* Currently in partial or full remission from a depressive or manic episode
* Under active clinical care

Inclusion Criteria for Adolescents:

* Speaks English or Spanish
* Presence of at least one current mood symptom meeting DSM-IV Criterion A and at least one depression or mania symptom meeting DSM-IV Criterion B
* Depression, irritability, anhedonia, or elated mood scored at level 2 or 3 on the KSADS-PL
* Mania symptom scored at level 2 or 3 on the KSADS-PL scale
* Score of less than 40 on the CDRS-R scale
* Score of less than 15 on the YMRS scale
* Mild-moderate functional impairment, defined as a score of greater than 61 and less than 75 on the C-GAS scale

Exclusion Criteria for Parents:

* History of psychosis within 1 month of study entry
* At risk for suicide within 1 month of study entry

Exclusion Criteria for Adolescents:

* Past major depressive or manic episode
* Current or past psychosis
* History of suicide attempts
* Current substance use disorder
* Use of psychotropic medications and other medications that might impact mood (e.g., steroids)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2006-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Verdeli, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates:10/06-5/10 Location: New York State Psychiatric Institute (mental health research and patient care)
Pre-assignment Details: Enrolled subjects were excluded from the trial because they were found to be either too symptomatic or asymptomatic
Groups:
- Interpersonal Psychotherapy for Prevention: Participants will receive 12 sessions of interpersonal psychotherapy for prevention of a mood disorder
- Educational Clinical Monitoring: Participants will receive educational clinical monitoring consisting of sessions of psychoeducation about mood disorders and monthly visits with a study therapist.
Period: Acute Phase
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Started | 2 | 5
Completed | 2 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow-up
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Started | 2 | 4
Completed | 1 | 1
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- IPT- Prevention for Adolescents: Participants will receive interpersonal psychotherapy for prevention with adolescents
  Interpersonal psychotherapy for prevention with adolescents: Individual interpersonal psychotherapy with the adolescents will be conducted over 12 weeks and will include a family psychoeducation component.
- Educational and Clinical Monitoring: Participants will receive educational clinical monitoring
  Educational clinical monitoring will include two individual sessions of psychoeducation on mood disorders with the adolescent followed by monthly (and if needed bimonthly) meetings with therapist. If more sessions are required, a referral will be made.
- Total: Total of all reporting groups
Arm/Group | IPT- Prevention for Adolescents | Educational and Clinical Monitoring | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 5 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: K SADS-Present Version (KSADS-P)
Description: A semi-structured interview designed to assess present episode of psychiatric illness according to DSM-IV criteria. The mood, anxiety, substance use and disruptive disorders sections were administered.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 2 | 4
participants
  Participants with sub-syndromal depression | 0 | 2
  Participants with sub-syndromal mania | 1 | 0
  Participants with current Oppositional defiant dis | 1 | 1
  Participants with current Depression | 0 | 1
  Participants with current Specific phobia | 1 | 0
  Participants with current subsyndromal PTSD | 0 | 1

2. Primary Outcome: K SADS-Present Version (KSADS-P)
Description: A semi-structured interview designed to assess present episode and episode since last assessment of psychiatric illness according to DSM-IV criteria. The mood, anxiety, substance use and disruptive disorders sections were administered.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 1 | 2
participants
  Participants with sub-syndromal depression | 0 | 1
  Participants with Specific phobia | 1 | 0
  Participant with major depression | 0 | 1

3. Primary Outcome: K SADS-Present Version (KSADS-P)
Description: as for outcome 2
Time Frame: 12 months
Population: At the 12 month follow up timepoint only 1 participant was available and willing to be assessed.
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 1
participants
  Participants with sub-syndromal depression |  | 1
  Participants with sub-syndromal mania |  | 1

4. Primary Outcome: K SADS-Present Version (KSADS-P)
Description: as for outcome 2
Time Frame: 18 months
Population: At the 18 month follow up point only 1 participant was available and willing be assessed.
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 0
participants
  Participants with sub-syndromal depression | 0 |
  Participant with specific phobia | 1 |

5. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R)
Description: CDRS-R Total score measures the presence and severity of depression in children/adolescents. The scale has 17 items scored on a 1-to-5 (3 items)- or 1-to-7 (14 items)-point scale. Total scores range from 17 to 113. Lower scores indicate lower depression, scores > 41 indicate mild-moderate depression.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 26.50 (7.78) | 28.75 (7.85)

6. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R)
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 1 | 2
units on a scale | 26 (0) | 29.5 (2.12)

7. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R)
Description: as for outcome 5
Time Frame: 12 months
Population: At the 12 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 1
units on a scale |  | 31 (0)

8. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R)
Description: as for outcome 5
Time Frame: 18 months
Population: At the 18 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 0
units on a scale | 25 (0) |

9. Primary Outcome: Children's Global Assessment Scale (C-GAS)
Description: C-GAS is a clinician-rated measure of overall severity of disturbance. A single assigned score ranging from 0 (most severe level of impairment) to 100 (absence of impairment) represents level of functional impairment.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 76 (1.41) | 70 (4.16)

10. Primary Outcome: Children's Global Assessment Scale (C-GAS)
Description: as for outcome 9
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 2
units on a scale | 81 (0) | 77.5 (3.54)

11. Primary Outcome: Children's Global Assessment Scale (C-GAS)
Description: as for outcome 9
Time Frame: 12 months
Population: At the 12 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 1
units on a scale |  | 79 (0)

12. Primary Outcome: Children's Global Assessment Scale (C-GAS)
Description: as for outcome 9
Time Frame: 18 months
Population: At the 18 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 0
units on a scale | 79 (0) |

13. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: An 11-item clinician-rated instrument for assessing the severity of manic episodes. 7 of the items are rated on a scale 0-4 and 4 are rated from 0-8. Total scores can range from 0-60, with higher scores indicating greater severity of symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 7 (8.49) | 4.5 (4.04)

14. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 13
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 2
units on a scale | 2 (0) | 3.5 (0.71)

15. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 13
Time Frame: 12 months
Population: At the 12 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 1
units on a scale |  | 6 (0)

16. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 13
Time Frame: 18 months
Population: At the 18 month time point 1 participant was available /willing to be assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 0
units on a scale | 3 (0) |

17. Secondary Outcome: Attitudes Toward Treatment Questionnaire
Description: A 4 item measure to evaluate attitudes towards: length of treatment, helpfulness of therapist, effects of participating in research, and additional services desired. Each item had 3 response options: 1.positive (or longer treatment) 2.neutral (or length just right) 3. negative (or shorter treatment). Scores are summed with potential range from 4-12. Lower number indicates more positive attitude
Time Frame: Measured at Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 6.50 (2.12) | 7.20 (1.48)

18. Secondary Outcome: Emotion Regulation Questionnaire
Description: A self report 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).Items 1, 3, 5, 7, 8, 10 make up the Cognitive Reappraisal facet (score is averaged, i.e., the score lies between 1 and 7), higher score indicates higher Cognitive reappraisal).
  Items 2, 4, 6, 9 make up the Expressive Suppression facet (score is averaged, i.e., the score lies between 1 and 7, higher score indicates higher Expressive Suppression).
Time Frame: Measured at Week 12
Population: Data were not collected for 6 and 12 month time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale
  Cognitive reappraisal | 4.5 (0.42) | 4.02 (0.91)
  Emotional suppression | 3.35 (0.64) | 4.62 (1.32)

19. Secondary Outcome: Emotion Regulation Questionnaire
Description: A self-report10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).Items 1, 3, 5, 7, 8, 10 make up the Cognitive Reappraisal facet (score is averaged, i.e., the score lies between 1 and 7), higher score indicates higher Cognitive reappraisal).
  Items 2, 4, 6, 9 make up the Expressive Suppression facet (score is averaged, i.e., the score lies between 1 and 7, higher score indicates higher Expressive Suppression).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 1 | 2
units on a scale
  Cognitive reappraisal | 4 (0) | 3.5 (0.71)
  Emotional suppression | 3 (0) | 4.5 (0.71)

20. Secondary Outcome: Emotion Regulation Questionnaire
Description: as for outcome 18
Time Frame: 12 months and 18 months
Population: At the 12 and 18 months time point no participant was willing to be assessed on this secondary outcome measure (had limited time for these assessment visits)
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Family Assessment Device
Description: The General Functioning scale, that assesses the overall health/pathology of the family, is used for the study. The 12 item scores are averaged to calculate the total score, which ranges from 1-4, with higher scores reflecting worse functioning
Time Frame: Measured at Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 2.3 (0.85) | 2.7 (0.51)

22. Secondary Outcome: Family History Screen
Description: A clinician-administered instrument to the adolescent' parent, designed to screen for mood, anxiety, and other disorders in parent's first-degree relatives (parents, spouse).
Time Frame: Measured at Week 1 (baseline)
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
participants
  Participants w/ parent'srelatives w/mood disorde | 2 | 4
  Participants w/ parent's relatives w/ anxiety | 2 | 3
  Participants w/ parents relatives w/substance use | 1 | 2

23. Secondary Outcome: Mood Disorder Questionnaire
Description: A self-report inventory for the participant' parent that screens for history of a manic or hypomanic syndrome by including 13 yes/no items. A score >7 indicate possible history of mania/hypomania (coded as 1), <7 indicates potential absence of mania/hypomania (coded as 0)
Time Frame: Week 1
Population: This measure reflects parental mood.expressed as number of participants whose parent with BDI or BDII endorsed > 7(1)
Measure: Number; unit: participants
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
participants | 2 | 4

24. Secondary Outcome: Patient Health Questionnaire
Description: The PHQ-9 is a depression screen, administered to the adolescents parents in this study. The PHQ-9 scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Scores can range from 0-27, with higher score indicating higher depression levels.
Time Frame: Measured at Week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 12 (2.8) | 14.5 (3.70)

25. Secondary Outcome: Social Adjustment Scale - Self Report for Adolescents
Description: (SAS-SR) for adolescents, a self-report instrument with 23 questions that fall into 4 major categories: school, friends, family, and dating. Patients rate themselves for the past 2 weeks and they can receive either a total score or a domain specific score. The total score is used here. Each item is scored 1-5, the total score is the average of the scores on each item, possible range of scores 1-5, higher scores indicating worse functioning.
Time Frame: Measured at Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 4
units on a scale | 1.9 (0.42) | 2.5 (0.57)

26. Secondary Outcome: Social Adjustment Scale - Self Report for Adolescents
Description: as for outcome 25
Time Frame: 12 months and 18 months
Population: as for outcome 20
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Social Rhythm Metric Short Form
Description: The Social Rhythm Metric Short Form (SRM-Short Form) measures habitual time at which 5 daily events occur in a person's life over a one-week interval: what time the adolescent gets out of bed, makes first contact with another person, starts school, has dinner, and goes to bed.
Time Frame: Measured at Week 12 and Months 6, 12, and 18 post-treatment
Population: Participants were not filling out form (it required documentation during the week) and reconstructing it in the meetings with the clinician proved to be too time consuming. Measure was withdrawn from the assessment battery
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Treatment Credibility Scale
Description: Treatment Credibility Questionnaire. Participant and parent's expectancy about the perceived benefit of treatment will be assessed following the first intervention session after the treatment rationale is given. Adolescents were asked to rate how logical the treatment seemed to them, how confident they were that it would be successful, and how confident they would be in recommending the treatment to a friend. A 0- to 2-point rating scale (0 = none, 1 = some, 2 = a lot) was used (range of possible overall score 0-6, higher score indicating higher treatment credibility)
Time Frame: Measured at Week 1
Population: An ECM participant did not fill out her form
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpersonal Psychotherapy-Prevention | Educational and Clinical Monitoring
Number analyzed (Participants) | 2 | 3
units on a scale | 4 (1.41) | 3.75 (0.96)

ADVERSE EVENTS:
Time Frame: 21 months
Groups:
- Interpersonal Psychotherapy for Prevention: Participants will receive interpersonal psychotherapy for prevention with adolescents
  Interpersonal psychotherapy for prevention with adolescents: Individual interpersonal psychotherapy with the adolescents will be conducted over 12 weeks and will include a family psychoeducation component.
- Educational Clinical Monitoring: Participants will receive educational clinical monitoring
  Educational clinical monitoring: Educational clinical monitoring will include two individual sessions of psychoeducation on mood disorders with the adolescent followed by monthly (and if needed bimonthly) meetings with therapist. If more sessions are required, a referral will be made.
Arm/Group | Interpersonal Psychotherapy for Prevention | Educational Clinical Monitoring
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5

LIMITATIONS AND CAVEATS:
Limitations include a very small sample size due to recruitment difficulty. In addition, participation with follow-up evaluations was poor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No